CLINICAL TRIAL: NCT03547388
Title: Gemäßigte Ganzkörperhyperthermie Bei Patienten Mit Rezidivierten Plattenepithelkarzinomen Der Kopf-Hals Region Nach Hochdosierter Vorbestrahlung: Pilotstudie Zur Beeinflussung Des Tumormikromilieus.
Brief Title: Moderate Whole Body Hyperthermia for Patients Undergoing Re-irradiation for Head and Neck Cancer -Influence on the Tumor Microenvironment
Acronym: GKH-TMM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Erwin Braun foundation (Unknown)
Responsible Party: Principal Investigator, Sebastian Zschaeck, MD, Principal Investigator, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EA2/047/18
Record Dates: First submitted 2018-03-27; First posted 2018-06-06 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Head and Neck Neoplasms; Recurrence Tumor
Keywords: head and neck squamous cell carcinoma; hyperthermia; hypoxia; 18f-fluoromisonidazole; positron emission tomography; FMISO; PET; whole body hyperthermia; local recurrence; lymph node recurrence; radiochemotherapy
MeSH Terms: conditions — Head and Neck Neoplasms; Recurrence; Squamous Cell Carcinoma of Head and Neck; Hyperthermia; Hypoxia

STUDY DESIGN:
Intervention Model Description: Phase I feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): Additional application of weekly moderate whole-body hyperthermia concurrent to re-irradiation plus chemotherapy
  Interventions: Device: Moderate whole body hyperthermia using water-filtered IR-A-radiation

INTERVENTIONS:
Device: Moderate whole body hyperthermia using water-filtered IR-A-radiation — four to six applications of whole Body hyperthermia concomitant to radiochemotherapy. Additional measurement of Perfusion and hypoxia by 18F-FMISO hypoxia PET and magnetic resonance Imaging
  Other Names: hypoxia imaging using 18f-fluoromisonidazole before radiochemotherapy and during second week of treatment

SUMMARY:
The aim of the study is to determine the feasibility and efficacy of moderate weekly whole Body hyperthermia Treatment during radiochemotherapy for pre-irradiated locally or regionally recurrent head and neck squamous cell carcinomas.

The Primary aim of the study is feasibility, defined as 80% of patients completing at least four applications of hyperthermia.

Secondary endpoints include an increase of Tumor Perfusion by the use of hyperthermia, measured by magnetic resonance Imaging during week two of Treatment and reduction of Tumor hypoxia, measured by hypoxia specific Positron emission tomography.

DETAILED DESCRIPTION:
Previously irradiated patients with loco/ loco-regional recurrent head and neck squamous cell carcinomas usually undergo re-irradiation. However prognosis of these patients is unfavourable, especially for non-human papilloma virus associated cancers. Moderate whole body hyperthermia will be performed by water-filtered IR-A-radiation using a Heckel-HT3000 device.

Preclinical data have indicated that moderate whole body hyperthermia decreases intratumoral interstitial fluid pressure and leads to increased perfusion of the tumor. The study investigates if this holds also true in patients and leads to a marked decrease of tumor hypoxia, measured by 18F-Fluoromisonidazole PET.

The Primary aim of the study is feasibility, defined as 80% of patients completing at least four applications of hyperthermia.

Secondary endpoints include an increase of Tumor Perfusion by the use of hyperthermia, measured by magnetic resonance Imaging during week two of Treatment and reduction of Tumor hypoxia, measured by hypoxia specific Positron emission tomography.

ELIGIBILITY:
Inclusion Criteria:

* patients with unresectable local, regional or loco-regional recurrent non HPV-associated squamous cell head and neck cancer with prior high-dose radiotherapy of the head and neck region
* time interval of 6 months to 5 years after completion of last radiotherapy of the head and neck region
* Completed staging examinations, preferentially 18f-fluorodeoxyglucose (FDG) PET of the whole body
* general health condition according to ECOG status of 0,1 or 2
* age between 18 and 75 years
* written informed consent

Exclusion Criteria:

* HPV associated primary tumor or recurrent tumor
* recurrence more than 5 years after end of previous radiotherapy
* Any medical circumstances impeding the application of radiotherapy, concomitant chemotherapy or whole body hyperthermia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2020-05-04 (Actual)

PRIMARY OUTCOMES:
feasibility of whole body hyperthermia as adjunct to radiochemotherapy | within 6 weeks of treatment with radiochemotherapy
  feasibility is defined as at least 4 cycles of whole body hyperthermia in 80% of patients

SECONDARY OUTCOMES:
Reduction of positron emission tomography (PET) measured hypoxia | 1 year (recruitment) plus additional 2 weeks (evaluation of PET parameter)
  defined as at least 80% reduction of the tumor to background ratio measured at the end of the second week of treatment compared to pre-treatment
magnetic resonance imaging (MRI) measured perfusion changes | 1 year (recruitment) plus additional 2 weeks (evaluation of MRI parameter)
  measured before treatment and at the end of week 2
Patient reported quality of life (head and neck cancer specific quality of life) | 3 years (i.e. recruitment plus two years of follow-up)
  measured by questionnaires according to EORTC (H&N35) and Transformation of absolute values to percentual values.
Patient reported quality of life (general quality of life) | 3 years (i.e. recruitment plus two years of follow-up)
  measured by questionnaires according to EORTC (C30) and Transformation of absolute values to percentual values.
Local control after 2 years of follow-up | 3 years (1 year recruitment, 2 years follow-up)
  From start of re-irradiation. Analysis will be performed by cox regression and log-rank analyses.
Loco-regional control after 2 years of follow-up | 3 years (1 year recruitment, 2 years follow-up)
  From start of re-irradiation. Analysis will be performed by cox regression and log-rank analyses.
Overall survival after 2 years of follow-up | 3 years (1 year recruitment, 2 years follow-up)
  From start of re-irradiation. Analysis will be performed by cox regression and log-rank analyses.
Freedom from distant metastases after 2 years of follow-up | 3 years (1 year recruitment, 2 years follow-up)
  From start of re-irradiation. Analysis will be performed by cox regression and log-rank analyses.
Tumor response | 1 year (recruitment) and 3 months (follow-up)
  Response of the irradiated tumor 3 months after end of treatment according to recist criteria

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Zschaeck, MD, Principal Investigator — Department of Radiation Oncology, Charité Universitätsmedizin Berlin, Augustenburger Platz 1, 13353, Berlin, Germany
Locations (1):
- Klinik für Radioonkologie und Strahlentherapie, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided
pseudonymized data may be shared upon reasonable request if accepted by all participating ethical commissions

REFERENCES:
- [Derived] Zschaeck S, Weingartner J, Ghadjar P, Wust P, Mehrhof F, Kalinauskaite G, Ehrhardt VH, Hartmann V, Tinhofer I, Heiland M, Coordes A, Kofla G, Budach V, Stromberger C, Beck M. Fever range whole body hyperthermia for re-irradiation of head and neck squamous cell carcinomas: Final results of a prospective study. Oral Oncol. 2021 May;116:105240. doi: 10.1016/j.oraloncology.2021.105240. Epub 2021 Feb 21. PMID 33626457